CLINICAL TRIAL: NCT03136952
Title: How Cerebral Oxygenation Correlates, Measured at Various Cranial Points, Frontally and Occipital in Children Under 1 Years Old, During General Anesthesia and Surgery
Brief Title: Cerebral Oxygenation, Different Measurement Points and Their Correlation in Pediatric Population
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Pether Jildenstal, Ass.professor, Göteborg University
Other Study IDs: Dnr 106-17.
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia Complication; Surgical Blood Loss
Keywords: NIRS; Monitoring; Pediatric
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric children under 1 yrs old: Observation study of two measurement points of cerebral oxygenation
  Interventions: Device: NIRS frontal and occipital

INTERVENTIONS:
Device: NIRS frontal and occipital — NIRS frontal and occipital on pediatric population during general anesthesia

SUMMARY:
Children who undergo surgery routinely for surgery that risk high levels of circulatory changes (eg heart surgery) is currently used routinely monitoring as regional oxygenation technology of the brain (NIRS). Near infrared spectroscopy (NIRS) is a technique for measuring regional oxygen saturation, indirect autoregulation of brain. We know that reduced oxygenation of the brain can occur with severe immediate blood loss. We in the research group has been able to note that in children who undergo surgery for cranioplasty interventions <1 year old, when they have ongoing excessive bleeding, decreases oxygenation in the brain and sometimes sharply before we can replace the loss of blood, even the blood pressure can be adequately maintained. Perioperative hypovolemia is a risk factor upset autoregulation of brain. Respect of which the mean arterial pressure (MAP) required to maintain intact autoregulation during general anesthesia still lacks a scientific consensus.

By illuminating the skin and underlying tissue with infrared light in the spectra of 700 to 1100nm, it is possible to measure regional oxygen saturation in various tissues. At cerebral measuring sensor is placed frontally, just below the hairline. INVOS then returns the absolute values of cerebral oxygen saturation frontally in the area where the sensor is placed.

A frontal placement may in some cases be impractical / impossible and thus limits the ability to monitor the brains of children with different types of surgery or body positions. At certain cranioplastic intervention surgery a frontal placement is not always possible, partly because of surgical technic reasons, but also that the child may have to lie prone during surgery. An alternative placement of INVOS sensor could mean greater opportunities to monitor cerebral oxygen saturation and thus increase patient safety within the mentioned categories of patients. An occipital location is practically possible in many cases. The purpose of this study is to investigate whether a occipital located sensor can measure cerebral oxygen saturation in a reliable manner.

DETAILED DESCRIPTION:
We want to study patients undergoing cleft lip and palate plastic surgery at Sahlgrenska University Hospital. This population has been chosen because it is an age group that is homogeneous and suits our aim "two different measuring points (frontal and occipitalt) of sensors for regional cerebral oxygenation in children under 1 yrs old, during general anesthesia and surgery. We will use a INVOS 5100 (the latest version of INVOS). A sensor will be applied, frontally and occipital on the head.

Patients will be enrolled consecutively when they have been planned for surgery, at Salhgrenska University Hospital.

Perioperative data will be registered in 5-minute intervals from frontally and occipital measurements. The measurements begin before the patient is anesthetized and ends when the patient is extubated.

All monitoring data during the general anesthesia will be obtained and documented in a data sheet.

ELIGIBILITY:
Inclusion Criteria:

- All children who will undergo cleft lip & palate surgery during general anesthesia.

Exclusion Criteria: Braintumor, neuropsychiatric diseases or ASA 3 classification.

-

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under one yrs old which shall undergo cleft lip & palate surgery during general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
NIRS correlation | 1 yr
  NIRS correlation between frontal and occipital measurement points

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska academy, University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No